CLINICAL TRIAL: NCT03819764
Title: Cost-effectiveness and Efficacy of a Combined Intervention to Facilitate Motor Recovery Following Stroke
Brief Title: Cost-effectiveness of Forced Aerobic Exercise for Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Susan Linder, Project Scientist, Principle Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-734
Record Dates: First submitted 2019-01-17; First posted 2019-01-29 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases
Keywords: stroke; aerobic exercise; forced exercise; repetitive task practice; arm function; upper extremity
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise & Repetitive Task Practice (Active Comparator): Participants will perform the following:
  1. 45 minutes of cycling
  2. 45 minutes of upper extremity repetitive arm exercises
  Interventions: Behavioral: Aerobic Exercise; Behavioral: Upper Extremity Repetitive Task Practice
- Upper Extremity Repetitive Task Practice Only (Active Comparator): Participants will perform the following:
  1. 90 minutes of upper extremity repetitive arm exercises
  Interventions: Behavioral: Upper Extremity Repetitive Task Practice

INTERVENTIONS:
Behavioral: Aerobic Exercise — Cycling on a recumbent stationary bike with a specialized motor that forces the individual to cycle approximately 30-35% faster than your self-selected speed
  Arms: Aerobic Exercise & Repetitive Task Practice
Behavioral: Upper Extremity Repetitive Task Practice — Repetitive arm exercises

SUMMARY:
The purpose of this study is to investigate whether aerobic exercise improves the participant's ability to recover function in the arm and leg affected by the participant's stroke. The investigators are also calculating the cost effectiveness of the rehabilitation interventions.

DETAILED DESCRIPTION:
The aims of the study are to determine the clinical efficacy and cost-effectiveness of combining aerobic exercise training with upper extremity motor task practice to improve motor recovery following stroke. It is hypothesized that the neurophysiologic impact of aerobic exercise may augment motor recovery associated with motor task practice. To test this hypothesize, 60 individuals with chronic stroke will be recruited to participate in this randomized clinical trial. Following screening and informed consent, all participants will undergo an exercise stress test to determine response to maximal exertion. Following the stress test, baseline clinical assessments will be obtained to quantify upper extremity function, gait, endurance, and self-reported quality of life. Additionally, variables to determine degree of disability will be obtained. Individuals will be randomized to one of two interventions: 45 min of forced-rate aerobic exercise paired with 45 min of upper limb repetitive task practice or two back-to-back 45-minute sessions of upper limb repetitive task practice. The interventions will occur 3 times per week for 8 weeks. Outcomes assessing motor function and disability will be repeated at mid-treatment, end of treatment, and at 4 weeks, 6-months and 12-months following end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 6 months following single ischemic or hemorrhagic stroke confirmed with neuroimaging,
2. Fugl-Meyer motor score 19-55 in the involved upper extremity,
3. Ambulatory ≥ 20 meters with no more than contact guard assistance, and
4. 18-85 years of age.

Exclusion Criteria:

1. hospitalization for myocardial infarction, heart failure or heart surgery within 3 months,
2. cardiac arrhythmia,
3. hypertrophic cardiomyopathy,
4. severe aortic stenosis,
5. pulmonary embolus,
6. significant contractures,
7. anti-spasticity injection within 3 months of enrollment and
8. other contraindication to exercise

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Linder, DPT, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Linder SM, Rilinger R, Learman K, Miller Koop M, Streicher M, Davidson S, Miller C, Harris D, Corrigan P, Bethoux F, Alberts JL. Forced-Rate Aerobic Cycling Improves Locomotor Function and Gait Biomechanics in Individuals With Chronic Stroke: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2025 Dec 1;104(12):1147-1154. doi: 10.1097/PHM.0000000000002785. Epub 2025 Jul 4. PMID 40720308
- [Derived] Linder SM, Bischof-Bockbrader A, Davidson S, Li Y, Lapin B, Singh T, Lee J, Bethoux F, Alberts JL. The Utilization of Forced-Rate Cycling to Facilitate Motor Recovery Following Stroke: A Randomized Clinical Trial. Neurorehabil Neural Repair. 2024 Apr;38(4):291-302. doi: 10.1177/15459683241233577. Epub 2024 Feb 29. PMID 38420848
- [Derived] Linder SM, Lee J, Bethoux F, Persson D, Bischof-Bockbrader A, Davidson S, Li Y, Lapin B, Roberts J, Troha A, Maag L, Singh T, Alberts JL. An 8-week Forced-rate Aerobic Cycling Program Improves Cardiorespiratory Fitness in Persons With Chronic Stroke: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2024 May;105(5):835-842. doi: 10.1016/j.apmr.2024.01.018. Epub 2024 Feb 11. PMID 38350494

RESULTS

PARTICIPANT FLOW:
Groups:
- Aerobic Exercise & Repetitive Task Practice: Participants will perform the following:
  1. 45 minutes of cycling
  2. 45 minutes of upper extremity repetitive arm exercises
  Aerobic Exercise: Cycling on a recumbent stationary bike with a specialized motor that forces the individual to cycle approximately 30-35% faster than self-selected speed
  Upper Extremity Repetitive Task Practice: Repetitive arm exercises
- Upper Extremity Repetitive Task Practice Only: Participants will perform the following:
  1. 90 minutes of upper extremity repetitive arm exercises
  Upper Extremity Repetitive Task Practice: Repetitive arm exercises
Period: Overall Study
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Started | 30 | 30
Completed | 29 | 27
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Aerobic Exercise & Repetitive Task Practice: Participants will perform the following:
  1. 45 minutes of cycling
  2. 45 minutes of upper extremity repetitive arm exercises
  Aerobic Exercise: Cycling on a recumbent stationary bike with a specialized motor that forces the individual to cycle approximately 30-35% faster than your self-selected speed
  Upper Extremity Repetitive Task Practice: Repetitive arm exercises
- Total: Total of all reporting groups
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (11.5) | 60.2 (9.8) | 60.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 29
  Male | 18 | 13 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 30 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 23 | 24 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Assessment (FMA)
Description: The Fugl-Meyer Assessment is a 33 item assessment of post-stroke upper extremity impairment. Total score is reported, scores range from 0-66, with higher scores indicating a better outcome.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
score on a scale | 32.5 (16.6) | 32.8 (18.6)

2. Primary Outcome: Fugl-Meyer Assessment (FMA)
Description: as for outcome 1
Time Frame: midpoint (4 weeks from Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
score on a scale | 44.0 (11.8) | 41.2 (13.4)

3. Primary Outcome: Fugl-Meyer Assessment (FMA)
Description: as for outcome 1
Time Frame: end of treatment (8 weeks from Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
score on a scale | 44.6 (12.5) | 42.1 (13.5)

4. Primary Outcome: Fugl-Meyer Assessment (FMA)
Description: as for outcome 1
Time Frame: end of treatment +4 weeks (12 weeks from Baseline)
Population: individuals with chronic stroke and residual upper limb paresis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
score on a scale | 44.6 (12.5) | 42.1 (13.5)

5. Primary Outcome: Fugl-Meyer Assessment (FMA)
Description: as for outcome 1
Time Frame: end of treatment +6 months (8 months from Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
score on a scale | 45.1 (12.8) | 43.7 (14.3)

6. Primary Outcome: Fugl-Meyer Assessment (FMA)
Description: as for outcome 1
Time Frame: end of treatment +1 year (14 months from Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
score on a scale | 44.8 (12.9) | 46.8 (13.6)

7. Primary Outcome: Action Research Arm Test (ARAT)
Description: The Action Research Arm Test is an assessment of post-stroke upper extremity function. Total score is reported, scores range from 0-57, with higher scores indicating a better outcome. The test includes 4 subscales: grasp (6 items, score range 0-18), grip (4 items, score range 0-12), pinch (6 items, score range 0-18), and gross motor (3 items, score range 0-9 ) which are added up for the total score. For all subscales, higher scores indicate better function.
Time Frame: Baseline
Population: individuals with chronic stroke and residual upper limb paresis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
score on a scale
  ARAT Total | 32.5 (16.6) | 32.8 (18.6)
  ARAT Grasp | 11.2 (5.7) | 11.4 (6.8)
  ARAT Grip | 6.8 (3.1) | 6.0 (3.9)
  ARAT Pinch | 8.0 (6.6) | 8.5 (7.0)
  ARAT Gross | 6.5 (2.3) | 6.9 (2.3)

8. Primary Outcome: Action Research Arm Test (ARAT)
Description: as for outcome 7
Time Frame: end of treatment (8 weeks from Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
score on a scale
  ARAT Total | 37.7 (17.9) | 36.4 (18.5)
  ARAT Grasp | 13.0 (6.2) | 12.6 (6.6)
  ARAT Grip | 7.6 (3.6) | 7.1 (4.0)
  ARAT Pinch | 9.9 (6.9) | 9.4 (7.1)
  ARAT Gross | 7.2 (2.4) | 7.3 (2.1)

9. Primary Outcome: Action Research Arm Test (ARAT)
Description: The Action Research Arm Test is an assessment of post-stroke upper extremity function. Total score is reported, scores range from 0-57, with higher scores indicating a better outcome.
Time Frame: end of treatment +4 weeks (12 weeks from Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
score on a scale
  ARAT Total | 39.3 (18.2) | 36.2 (19.8)
  ARAT Grasp | 13.7 (6.0) | 12.6 (6.8)
  ARAT Grip | 7.8 (4.1) | 7.0 (4.4)
  ARAT Pinch | 10.4 (7.1) | 9.4 (7.3)
  ARAT Gross | 7.4 (2.4) | 7.2 (2.41)

10. Primary Outcome: Action Research Arm Test (ARAT)
Description: as for outcome 7
Time Frame: end of treatment +6 months (8 months from Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
score on a scale
  ARAT Total | 37.1 (19.4) | 39.1 (18.3)
  ARAT Grasp | 13.2 (6.4) | 13.6 (6.6)
  ARAT Grip | 7.5 (4.2) | 7.4 (4.2)
  ARAT Pinch | 9.1 (7.8) | 10.2 (7.2)
  ARAT Gross | 7.2 (2.5) | 8.0 (1.7)

11. Primary Outcome: Action Research Arm Test (ARAT)
Description: as for outcome 7
Time Frame: end of treatment +1 year (14 months from Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
score on a scale
  ARAT Total | 38.5 (18.4) | 40.9 (17.6)
  ARAT Grasp | 14.2 (6.0) | 14.1 (6.3)
  ARAT Grip | 7.1 (4.0) | 8.0 (4.1)
  ARAT Pinch | 10.0 (7.5) | 10.7 (7.2)
  ARAT Gross | 7.3 (2.5) | 8.0 (1.6)

12. Secondary Outcome: Wolf Motor Function Test (WMFT)
Description: The Wolf Motor Function Test includes 15 timed tasks for the affected upper extremity. Times for timed tasks are transformed and reported as geometric mean (standard deviation). Lower times indicate better performance.
Time Frame: Baseline
Population: individuals with chronic stroke with residual upper limb paresis
Measure: Geometric Mean (Standard Deviation); unit: time in seconds
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
time in seconds | 11.0 (3.0) | 14.9 (3.3)

13. Secondary Outcome: Stroke Impact Scale (SIS)
Description: The Stroke Impact Scale is a self-reported questionnaire evaluating quality of life. 8 domains are assessed including: physical problems, memory and thinking, feelings, communication, activities of daily living (ADLs), mobility, hand use, and meaningful activities. Scores for all domains are normalized and range from 0-100, with higher scores indicating a better self-perceived quality of life. The last domain (stroke recovery) asks the individual to rate their recovery on a scale of 0-100, with 0 indicating no recovery and 100 indicating full recovery.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
score on a scale
  SIS Physical Problem | 50.6 (17.1) | 47.8 (19.4)
  SIS Memory and Thinking | 86.5 (13.4) | 83.7 (16.4)
  SIS Feelings | 80.0 (14.4) | 69.8 (18.7)
  SIS Communication | 87.2 (19.4) | 83.9 (18.8)
  SIS ADL's | 73.4 (14.5) | 67.8 (18.8)
  SIS Mobility | 81.5 (12.9) | 75.9 (17.7)
  SIS Hand Use | 41.9 (27.2) | 42.5 (28.9)
  SIS Meaningful Activities | 61.4 (23.8) | 63.0 (25.8)
  SIS Stroke Recovery Score | 62.3 (20.8) | 52.5 (23.3)

14. Secondary Outcome: Stroke Impact Scale (SIS)
Description: as for outcome 13
Time Frame: end of treatment (8 weeks from Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
score on a scale
  SIS Physical Problem | 58.4 (14.9) | 54.8 (22.6)
  SIS Memory and Thinking | 88.3 (14.8) | 83.7 (19.9)
  SIS Feelings | 81.6 (14.2) | 77.6 (16.5)
  SIS Communication | 87.6 (17.6) | 88.9 (17.2)
  SIS ADLs | 76.9 (13.8) | 74.4 (16.2)
  SIS Mobility | 84.4 (12.7) | 78.3 (18.2)
  SIS Hand Use | 54.5 (26.4) | 52.6 (26.3)
  SIS Meaningful Activities | 73.8 (19.0) | 69.8 (17.7)
  SIS Stroke Recovery | 64.6 (19.4) | 63.4 (19.8)

15. Secondary Outcome: Stroke Impact Scale (SIS)
Description: as for outcome 13
Time Frame: end of treatment +6 months (8 months from Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
score on a scale
  SIS Physical Problem | 60.8 (20.2) | 54.9 (22.3)
  SIS Memory and Thinking | 87.3 (15.1) | 85.3 (15.2)
  SIS Feelings | 83.5 (12.7) | 79.5 (15.1)
  SIS Communication | 89.9 (15.6) | 91.0 (11.0)
  SIS ADL's | 77.0 (15.4) | 77.9 (13.7)
  SIS Mobility | 84.6 (13.3) | 80.8 (14.4)
  SIS Hand Use | 50.5 (27.8) | 52.6 (26.7)
  SIS Meaningful Activities | 75.0 (17.4) | 67.6 (20.3)
  SIS Stroke Recovery Score | 68.0 (17.7) | 66.5 (21.5)

16. Secondary Outcome: Stroke Impact Scale (SIS)
Description: as for outcome 13
Time Frame: end of treatment +1 year (14 months from Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
score on a scale
  SIS Physical Problem | 60.1 (22.1) | 59.4 (19.7)
  SIS Memory and Thinking | 88.1 (16.6) | 90.9 (11.6)
  SIS Feelings | 82.5 (16.8) | 81.5 (14.1)
  SIS Communication | 88.8 (19.2) | 91.2 (10.7)
  SIS ADL'S | 74.5 (16.1) | 77.0 (14.4)
  SIS Mobility | 83.3 (12.6) | 84.3 (12.3)
  SIS Hand Use | 49.0 (28.1) | 52.8 (24.9)
  SIS Meaningful Activities | 69.3 (26.9) | 73.0 (19.2)
  SIS Stroke Recovery Score | 65.7 (20.6) | 66.9 (22.8)

17. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS-29)
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS-29) is a self-reported questionnaire evaluating physical, mental, and social health. T-scores are reported separately for Anxiety, Depression, Fatigue, Sleep Disturbance, Ability to Participate in Social Roles and Activities, Physical Function, and Pain Interference.
  * A score of 50 represents the population mean.
  * A score of 40 is one standard deviation lower than the mean of the reference population.
  * A score of 60 is one standard deviation higher than the mean of the reference population.
  * For PROMIS measures, higher scores for domains measuring symptoms is indicative of greater symptom burden. Therefore, higher scores are worse for fatigue, anxiety, depression, sleep disturbance, and pain interference. For the domains of Physical Function and Participation, higher scores indicate better function and better participation, respectively.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
T-score
  Physical | 39.6 (6.6) | 40.1 (5.8)
  Anxiety | 49.7 (8.1) | 49.9 (8.3)
  Depression | 49.2 (7.9) | 48.9 (7.6)
  Fatigue | 47.8 (8.7) | 48.0 (8.6)
  Sleep Disturbance | 46.8 (9.9) | 45.5 (9.9)
  Participation | 46.3 (8.4) | 45.8 (8.5)
  Pain Interference | 49.0 (8.5) | 47.4 (6.9)

18. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS-29)
Description: as for outcome 17
Time Frame: end of treatment (8 weeks from Baseline)
Population: individuals with chronic stroke and residual upper limb paresis
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
T-score
  Physical | 40.8 (6.5) | 41.3 (5.3)
  Anxiety | 48.8 (9.4) | 48.2 (9.8)
  Depression | 49.6 (8.6) | 49.2 (8.7)
  Fatigue | 48.5 (8.7) | 47.1 (8.9)
  Sleep Disturbance | 46.2 (9.0) | 44.7 (8.3)
  Participation | 49.3 (9.1) | 49.9 (9.7)
  Pain Interference | 49.7 (8.8) | 48.2 (8.5)

19. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS-29)
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS-29) is a self-reported questionnaire evaluating physical, mental, and social health. T-scores are reported separately for Anxiety, Depression, Fatigue, Sleep Disturbance, Ability to Participate in Social Roles and Activities, Physical Function, and Pain Interference.
  * A score of 50 represents the population mean.
  * A score of 40 is one standard deviation lower than the mean of the reference population.
  * A score of 60 is one standard deviation higher than the mean of the reference population.
  * For PROMIS measures, higher scores for domains measuring symptoms is indicative of greater symptom burden. Therefore, higher scores are worse for fatigue, anxiety, depression, sleep disturbance, and pain interference. For the domains of Physical Function and Participation, higher scores indicate better function and better participation, respectively.easured.
Time Frame: end of treatment +6 months (8 months from Baseline)
Population: individuals with chronic stroke and residual upper limb paresis
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
T-score
  Physical | 42.0 (7.6) | 41.4 (7.4)
  Anxiety | 47.5 (9.0) | 47.6 (9.0)
  Depression | 48.3 (7.6) | 47.6 (7.4)
  Fatigue | 47.1 (9.8) | 45.3 (10.2)
  Sleep Disturbance | 45.2 (8.9) | 44.5 (10.7)
  Participation | 51.0 (9.7) | 51.5 (10.9)
  Pain Interference | 51.3 (8.0) | 50.0 (8.4)

20. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS-29)
Description: as for outcome 17
Time Frame: end of treatment +1 year (14 months from Baseline)
Population: individuals with chronic stroke and residual upper limb paresis
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
T-score
  Physical | 41.1 (6.8) | 40.5 (5.9)
  Anxiety | 47.9 (9.7) | 49.1 (10.4)
  Depression | 48.2 (8.6) | 48.1 (9.2)
  Fatigue | 46.8 (8.6) | 47.7 (9.3)
  Sleep Disturbance | 45.2 (9.7) | 43.6 (10.4)
  Participation | 49.6 (9.2) | 48.4 (10.1)
  Pain Interference | 49.4 (8.6) | 49.4 (9.2)

21. Secondary Outcome: Center for Epidemiological Studies-Depression (CES-D)
Description: The Center for Epidemiological Studies-Depression (CES-D) is a 20 item assessment of depressive symptomology. Total score is reported, scores range from 0-60, with higher scores indicating higher risk of depression. A score of 16 or more is indicative of depression.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
units on a scale | 11.3 (8.5) | 9.6 (7.4)

22. Secondary Outcome: Center for Epidemiological Studies-Depression (CES-D)
Description: as for outcome 21
Time Frame: end of treatment (8 weeks from Baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
units on a scale | 9.9 (9.3) | 8.8 (9.3)

23. Secondary Outcome: Center for Epidemiological Studies-Depression (CES-D)
Description: as for outcome 21
Time Frame: end of treatment +6 months (8 months from Baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
units on a scale | 9.3 (7.8) | 8.6 (8.5)

24. Secondary Outcome: Center for Epidemiological Studies-Depression (CES-D)
Description: as for outcome 21
Time Frame: end of treatment +1 year (14 months from Baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
units on a scale | 9.3 (8.3) | 9.7 (9.7)

25. Secondary Outcome: Six-Minute Walk Test (6MWT)
Description: The Six-Minute Walk Test (6MWT) measures total distance traveled over a 6 minute period.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: Meters
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
Meters | 264.4 (118.4) | 285.5 (160.3)

26. Secondary Outcome: Six-Minute Walk Test (6MWT)
Description: The Six-Minute Walk Test (6MWT) measures total distance traveled over a 6 minute period.
Time Frame: end of treatment (8 weeks)
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
Meters | 327.1 (141.2) | 316.9 (170.0)

27. Secondary Outcome: Six-Minute Walk Test (6MWT)
Description: The Six-Minute Walk Test (6MWT) measures total distance traveled over a 6 minute period.
Time Frame: end of treatment +4 weeks (12 weeks from Baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
units on a scale | 339.3 (156.7) | 315.1 (170.5)

28. Secondary Outcome: Six-Minute Walk Test (6MWT)
Description: The Six-Minute Walk Test (6MWT) measures total distance traveled over a 6 minute period.
Time Frame: end of treatment +6 months (8 months from Baseline)
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
Meters | 339.3 (156.7) | 315.1 (170.5)

29. Secondary Outcome: Six-Minute Walk Test (6MWT)
Description: The Six-Minute Walk Test (6MWT) measures total distance traveled over a 6 minute period.
Time Frame: end of treatment +1 year (14 months from Baseline)
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
Meters | 320.8 (166.5) | 336.7 (170.3)

30. Secondary Outcome: Paretic Step Length
Description: Mean Paretic step length (cm) across two 2-minute walking trials
Time Frame: Baseline
Population: individuals with chronic stroke and residual hemiparesis who opted to have biomechanical gait assessment completed. This was a secondary outcome and included a subset of the total sample.
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 25 | 20
Centimeters | 40.4 (14.1) | 45.6 (12.7)

31. Secondary Outcome: Non-Paretic Step Length
Description: Mean Non-Paretic step length (cm) across two 2-minute walking trials
Time Frame: Baseline
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 25 | 20
Centimeters | 40.1 (15.5) | 44.2 (14.9)

32. Secondary Outcome: Paretic Step Length
Description: Mean Paretic step length (cm) across two 2-minute walking trials
Time Frame: end of treatment (8 weeks from Baseline)
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 25 | 20
Centimeters | 45.0 (12.6) | 46.9 (11.5)

33. Secondary Outcome: Non-Paretic Step Length
Description: Mean Non-Paretic step length (cm) across two 2-minute walking trials
Time Frame: end of treatment (8 weeks from Baseline)
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 25 | 30
Centimeters | 45.0 (15.3) | 46.1 (11.5)

34. Secondary Outcome: Non-Paretic Single Limb Percentage
Description: Percentage of gait cycle spent in single limb support
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 25 | 20
Percent | 29.1 (4.79) | 30.1 (2.64)

35. Secondary Outcome: Non-Paretic Single Limb Percentage
Description: Mean percentage of gait cycle spent in stance phase on the Non-Paretic lower extremity across two 2-minute walking trials
Time Frame: end of treatment (8 weeks from Baseline)
Population: individuals with chronic stroke and residual upper limb paresis who opted to have biomechanical gait assessment completed. This was a secondary outcome and included a subset of the total sample.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 25 | 20
Percent | 29.8 (4.73) | 30.5 (2.30)

36. Secondary Outcome: Modified Rankin Scale
Description: The modified Rankin Scale is a global outcome on a scale of 0-6 used to assess the degree of disability in patients with stroke as follows:
  0 No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
score on a scale | 2 [1 to 3] | 2 [1 to 3]

37. Secondary Outcome: Modified Rankin Scale
Description: as for outcome 36
Time Frame: end of treatment (8 weeks from Baseline)
Population: individuals with chronic stroke and residual hemiparesis
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
score on a scale | 2 [1 to 3] | 2 [1 to 3]

38. Secondary Outcome: Walking Cadence
Description: Steps walked per minute during two 2-minute walking trials
Time Frame: Baseline
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: steps/min
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 25 | 25
steps/min | 82.1 (17.2) | 86.1 (17.3)

39. Secondary Outcome: Walking Cadence
Description: Steps walked per minute during two 2-minute walking trials
Time Frame: end of treatment (8 weeks from Baseline)
Measure: Mean (Standard Deviation); unit: steps/min
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 25 | 20
steps/min | 86.1 (17.3) | 85.8 (15.4)

40. Secondary Outcome: Paretic Single Limb Percentage
Description: Percentage of gait cycle spent in single limb support
Time Frame: Baseline
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 25 | 20
Percentage | 26.8 (3.88) | 28.6 (2.76)

41. Secondary Outcome: Paretic Single Limb Percentage
Description: Percentage of gait cycle spent in single limb support
Time Frame: end of treatment (8 weeks from Baseline)
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 25 | 20
Percent | 27.9 (3.40) | 28.9 (2.70)

42. Secondary Outcome: Paretic Knee Range of Motion
Description: Mean peak degree of paretic knee flexion across two 2-minute walking trials
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 25 | 20
Degrees | 43.0 (16.9) | 54.1 (14.4)

43. Secondary Outcome: Paretic Knee Range of Motion
Description: Mean peak degree of paretic knee flexion across two 2-minute walking trials
Time Frame: end of treatment (8 weeks from Baseline)
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 25 | 20
Degrees | 44.0 (17.5) | 53.4 (12.5)

44. Secondary Outcome: Non-Paretic Knee Range of Motion
Description: Mean peak degree of non-paretic knee flexion across two 2-minute walking trials
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 25 | 20
Degrees | 53.6 (11.85) | 60.5 (9.12)

45. Secondary Outcome: Non-Paretic Knee Range of Motion
Description: Mean peak degree of non-paretic knee flexion across two 2-minute walking trials
Time Frame: end of treatment (8 weeks from Baseline)
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 25 | 20
Degrees | 54.8 (10.9) | 62.4 (6.41)

46. Secondary Outcome: Paretic Ankle Range of Motion
Description: Mean peak degree of paretic ankle dorsiflexion across two 2-minute walking trials
Time Frame: Baseline
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 25 | 20
Degrees | 17.8 (5.38) | 19.5 (6.45)

47. Secondary Outcome: Paretic Ankle Range of Motion
Description: Mean peak degree of paretic ankle dorsiflexion across two 2-minute walking trials
Time Frame: end of treatment (8 weeks from Baseline)
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 25 | 20
Degrees | 19.1 (5.46) | 19.1 (6.10)

48. Secondary Outcome: Non-Paretic Ankle Range of Motion
Description: Non-Paretic peak degree of non-paretic dorsiflexion across two 2-minute walking trials
Time Frame: Baseline
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 25 | 20
Degrees | 23.3 (8.74) | 23.7 (7.28)

49. Secondary Outcome: Non-Paretic Ankle Range of Motion
Description: Mean peak degree of non-paretic ankle dorsiflexion across two 2-minute walking trials
Time Frame: end of treatment (8 weeks from Baseline)
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 25 | 20
Degrees | 24.8 (8.48) | 23.2 (6.89)

50. Secondary Outcome: Paretic Hip Range of Motion (Sagittal Plane)
Description: Mean peak degree of paretic hip flexion across two 2-minute walking trials
Time Frame: Baseline
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 25 | 20
Degrees | 33.2 (9.39) | 37.4 (10.4)

51. Secondary Outcome: Paretic Hip Range of Motion (Sagittal Plane)
Description: Mean peak degree of paretic hip flexion across two 2-minute walking trials
Time Frame: end of treatment (8 weeks from Baseline)
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 25 | 20
Degrees | 35.6 (10.0) | 39.5 (7.64)

52. Secondary Outcome: Non-Paretic Hip Range of Motion (Sagittal Plane)
Description: Mean peak degree of non-paretic hip flexion across two 2-minute walking trials
Time Frame: Baseline
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 25 | 20
Degrees | 36.9 (9.35) | 41.3 (6.14)

53. Secondary Outcome: Non-Paretic Hip Range of Motion (Sagittal Plane)
Description: Mean peak degree of non-paretic hip flexion across two 2-minute walking trials
Time Frame: end of treatment (8 weeks from Baseline)
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 25 | 20
Degrees | 39.9 (9.37) | 43.0 (5.89)

54. Secondary Outcome: Wolf Motor Function Test (WMFT) Functional Ability Score
Description: The Wolf Motor Function Test Functional Ability Score quantifies movement quality. Scores range from 0-75, with higher scores indicating a better outcome.
Time Frame: End of Treatment (8 weeks from baseline)
Population: individuals with chronic stroke with residual upper limb paresis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
score on a scale | 3.4 (1.3) | 3.2 (1.4)

55. Secondary Outcome: Wolf Motor Function Test (WMFT) Grip Strength
Description: The Wolf Motor Function Test includes Grip strength measured by dynamometer
Time Frame: End of Treatment (8 weeks from baseline)
Population: individuals with chronic stroke with residual upper limb paresis
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
kg | 14.2 (8.5) | 14.1 (9.0)

56. Secondary Outcome: Wolf Motor Function Test (WMFT) Weight to Box
Description: The Wolf Motor Function Test includes the amount of weight the individual can lift onto a box using a wrist cuff weight ranging from 1-20 pounds. Higher indicates greater strength.
Time Frame: End of Treatment (8 weeks from baseline)
Population: individuals with chronic stroke with residual upper limb paresis
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
pounds | 10.6 (7.0) | 10.8 (7.2)

57. Secondary Outcome: Wolf Motor Function Test (WMFT)
Description: as for outcome 12
Time Frame: end of treatment (8 weeks from baseline)
Population: individuals with chronic stroke with residual upper limb paresis
Measure: Geometric Mean (Standard Deviation); unit: time in seconds
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
time in seconds | 8.2 (3.3) | 10.0 (3.7)

58. Secondary Outcome: Wolf Motor Function Test (WMFT) Functional Ability Score
Description: The WMFT Functional Ability Score quantifies movement quality. Scores range from 0-75, with higher scores indicating a better outcome.
Time Frame: Baseline
Population: individuals with chronic stroke with residual upper limb paresis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
score on a scale | 2.4 (1.1) | 2.7 (1.2)

59. Secondary Outcome: Wolf Motor Function Test (WMFT) Grip Strength
Description: The Wolf Motor Function Test includes Grip strength measured by dynamometer
Time Frame: baseline
Population: individuals with chronic stroke with residual upper limb paresis
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
kg | 13.8 (7.9) | 13.8 (8.9)

60. Secondary Outcome: Wolf Motor Function Test (WMFT) Weight to Box
Description: as for outcome 56
Time Frame: baseline
Population: individuals with chronic stroke with residual upper limb paresis
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
pounds | 8.2 (6.3) | 8.7 (7.2)

61. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS-29) Pain Intensity
Description: The Patient-Reported Outcomes Measurement Information System includes pain rated on a 0-10 scale with higher scores indicative of greater pain.
Time Frame: End of Treatment (8 weeks following baseline)
Population: individuals with chronic stroke and residual upper limb paresis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
units on a scale | 2.3 (2.6) | 2.6 (2.4)

62. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS-29) Pain Intensity
Description: The Patient-Reported Outcomes Measurement Information System includes pain rated rated on a 0-10 scale with higher scores indicative of greater pain.
Time Frame: Baseline
Population: individuals with chronic stroke and residual upper limb paresis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
units on a scale | 2.4 (2.1) | 2.4 (2.3)

63. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS-29) Pain Intensity
Description: as for outcome 61
Time Frame: end of treatment + 6 months (8 months from baseline)
Population: individuals with chronic stroke and residual upper limb paresis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
units on a scale | 2.3 (2.1) | 2.4 (2.0)

64. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS-29) Pain Intensity
Description: as for outcome 61
Time Frame: end of treatment + 12 months (14 months from baseline)
Population: individuals with chronic stroke and residual upper limb paresis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
Number analyzed (Participants) | 30 | 30
units on a scale | 2.7 (2.8) | 2.7 (2.3)

ADVERSE EVENTS:
Time Frame: Adverse experiences were collected up to 2 years from the start to the completion of the study.
Arm/Group | Aerobic Exercise & Repetitive Task Practice | Upper Extremity Repetitive Task Practice Only
All-Cause Mortality (participants affected / at risk) | 0/30 | 1/30
Serious Adverse Events (participants affected / at risk) | 2/30 | 2/30
Other Adverse Events (participants affected / at risk) | 5/30 | 8/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerobic Exercise & Repetitive Task Practice (N=30) | Upper Extremity Repetitive Task Practice Only (N=30)
Cancer Diagnosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) — patient diagnosed with prostate cancer 3 months following completion of intervention, unrelated to study intervention. He was unable to complete 6- and 12-month follow up assessments
Sepsis (Infections and infestations) | 0 (0) | 1 (1) — patient was being treated for skin cancer & lesion became infected;
Stroke (Vascular disorders) | 1 (1) | 1 (1) — one individual had recurrent stroke 6 months following completion of study while still enrolled in 1-year follow up
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerobic Exercise & Repetitive Task Practice (N=30) | Upper Extremity Repetitive Task Practice Only (N=30)
Skin Injury (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (3) | 8 (13)
Leg Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT03819764/Prot_SAP_001.pdf
  • Informed Consent Form (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT03819764/ICF_002.pdf